CLINICAL TRIAL: NCT06608121
Title: Study for the Development and Evaluation of Personalised Muscle Effort Generation Models for Patients With Upper Limb Motor Deficits
Brief Title: Upper Limb Muscle Strength Models for Patients With Motor Impairment.
Acronym: MusMapS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pôle Saint Hélier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2024-A01007-40
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Stroke; Multiple Sclerosis; Spinal Cord Injuries
Keywords: muscle strength; modeling; upper limb; motor impairment
MeSH Terms: conditions — Stroke; Multiple Sclerosis; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental)
  Interventions: Other: Upper limb isokinetic forces measurements

INTERVENTIONS:
Other: Upper limb isokinetic forces measurements — The trial is a single-center prospective interventional study. Patients aged 18 to 85 years hospitalized in a French rehabilitation center for stroke, multiple sclerosis or traumatic tetraplegia and presenting a motor deficit ≤3/5 at the shoulder and elbow will be included. MVF measurements will be performed using an isokinetic ergometer during a single session. Concentric and eccentric MVF, as well as the forces generated during passive motion, will be measured in shoulder external-internal rotation and in elbow flexion-extension, in the seated position. The demographic, anthropometric and medical data required for the study will be extracted from medical records. Patients' residual muscle strength will be described and modeled. Explanatory factors for model quality will be determined.

SUMMARY:
Upper limb motor impairments are common. They affect quality of life and can lead to dependency. They are mainly due to neurological conditions such as stroke, multiple sclerosis, and traumatic spinal cord injury. However, the contractile properties of muscle, in particular the maximum force that can be generated voluntarily (MVF) depending on joint angle and motion speed, have been mainly studied and modeled in healthy people. This study aims at developing mathematical models describing residual muscle forces in patients with motor impairments. The knowledge could guide patients' rehabilitation and could be useful for the development of robotic assistance systems that use patients' residual capacities to control the level of assistance provided.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 85
* A patient who is a member or beneficiary of a social security scheme
* Patients hospitalised at the Saint-Hélier rehabilitation centre for a stroke more than 15 days old, MS or SCI
* Patients with a motor deficit ≤3/5 on the MRC (Medical Research Council) scale in both internal-external shoulder rotation and elbow flexion-extension.
* Patient with voluntary consent to participate in this study.

Exclusion Criteria:

* Spasticity >3/4 on the Aschworth scale in the shoulder abductor or elbow flexor muscles.
* Cognitive impairment that may interfere with measurements (MOCA < 20/30)
* Presence of a pressure sore > stage 2 at the ischial level
* Recent trauma to limbs or spine
* Decompensated heart disease or other unbalanced pathology which contraindicates or may hinder isokinetic testing.
* Persons deprived of their liberty by a judicial or administrative decision
* Pregnant women, women in labour or nursing mothers.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2025-10-22 (Actual)

PRIMARY OUTCOMES:
Description of the residuals of the effort generation models, defined as the difference between the actual effort values and the modelled values: o Average residual of the models (mean ± standard deviation) (Main Evaluation Criterion) | From enrollment to the end of the participation at maximum 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Saint-Hélier, Rennes, France

IPD SHARING:
Plan to Share IPD: Undecided